CLINICAL TRIAL: NCT02569047
Title: ART and Hall Technique for the Management of Occlusal-proximal Caries in Primary Molars: A Randomized Clinical Trial
Brief Title: ART and Hall Technique for Management of Occlusal-proximal Caries in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: University of Dundee (Other); Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associated Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALLART
Record Dates: First submitted 2015-09-28; First posted 2015-10-06 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Dental Caries
Keywords: Atraumatic Restorative Treatment; Occlusoproximal; Primary Teeth; Glass Ionomer Cements; Hall Technique
MeSH Terms: conditions — Dental Caries | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atraumatic Restorative Treatment (Active Comparator): The cavity will be prepared according to the ART (Atraumatic Restorative Treatments) steps and filled with the dental material Glass Ionomer Cement without local anesthesia.
  Interventions: Procedure: Atraumatic Restorative Treatment
- Hall Technique (Experimental): The cavity will not receive any preparation. A stainless crown will be placed and cemented with the dental material Glass Ionomer Cement without local anesthesia.
  Interventions: Procedure: Hall Technique

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment — No local anaesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with Glass Ionomer Cement (GIC).The cavity will be filled with GIC. After the press-finger technique, the excess of material will be removed.
  Other Names: Equia Forte
  Arms: Atraumatic Restorative Treatment
Procedure: Hall Technique — It employs the cementation of preformed metal crowns (PMC) without the need of any prior teeth preparation or caries removal. No local anesthesia is used neither tooth preparation.Different sizes of PMCs will be tested until the smallest size that perfectly fit the tooth is achieved. The PMC will be loaded with the dental material glass ionomer cement (GIC) and placed. Child will asked to bite firmly on it, until it is fitted. The excess of GIC will be removed with hand instruments and dental floss.
  Other Names: Metal Crowns
  Arms: Hall Technique

SUMMARY:
The aim of this, two-arm, parallel group, patient-randomised controlled, superiority trial is to evaluate the survival rate of approximal Atraumatic Restorative Treatment (ART) restorations compared to the Hall Technique (HT) placed in a school setting. The investigators will recruit 120 schoolchildren (5-10 years) with at least one occlusal-proximal carious lesion in primary molar. They will be randomized and treated following best-practice protocols to either receive an ART restoration using the high-viscosity glass ionomer cement (EQUIA Forte, capsules, GC Corp.) or a preformed metal crown placed using the HT (3M ESPE) cemented with glass ionomer luting cement (Fuji I Capsules, GC Corp.). Baseline measures and outcome data (at reviews over a three year period) will be assessed through participant report, clinical examination and parent report/ questionnaires.

DETAILED DESCRIPTION:
The selected children will be randomly allocated into 2 groups. The control group will comprise cavities treated by ART, following the protocol proposed by Frencken and Holmgren (1999), while the experimental group will comprise cavities treated by HT, according to the guideline published by Innes and Evans (2011). The allocation of patients in each group will be carried out by a random list generated by a specific computer program. To ensure the allocation concealment, the sequence generated by randomization will be distributed in opaque, sealed envelopes, which will be opened by the operator during the treatment, only after the patient is ready to receive treatment.

Operators will be two undergraduate students in dentistry and one experienced specialist in pediatric dentistry that will be trained on how to prepare and fill the cavities according to the original procedures of ART (Frencken and Holmgren, 1999) and also according to HT (Innes and Evans, 2011). The training will include a lecture about the techniques used in this study, as well as a workshop held in the laboratory for students to train handling and application of treatments to be tested. They will also undergo a week of training with patients, to apply the different techniques before starting the study, the latter phase held at the Faculty of Dentistry, University of São Paulo, under the supervision of an experienced dentist in ART and HT.

Each child will be allocated for one of the operators with the aid of a random list. All treatments will be performed on the school premises, in field conditions without the use of dental chair or other facilities from a clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 5 and 10 years
* cooperative behavior
* presenting good health conditions
* whose parents or legal guardians accept and sign the consent form
* with at least one occluso-proximal lesion in primary molar
* only occlusal-proximal surfaces with caries lesions with dentin involvement
* cavities accessible to hand instruments used in ART
* absence of fistula or abscess near the selected tooth
* absence of pulp exposure in the selected tooth
* absence of mobility in the selected tooth
* cavity size in the selected tooth not be bigger than 2.0 mm in the mesial-distal and 2.5 in the occlusal-cervical and bucco-lingual directions.

Exclusion Criteria:

* children younger than 5 years and older than 10
* non-cooperative behavior
* without good health conditions
* whose parents or legal guardians did not accepted and signed the consent form
* without any occluso-proximal lesion in primary molar
* caries in the selected tooth reaching other surfaces (than occlusal-proximal surface)
* occlusal-proximal surface with caries without dentin involvement
* cavities not accessible to hand instruments
* fistula or abscess near the selected tooth
* pulp exposure in the selected tooth
* mobility in the selected tooth
* cavity size bigger than 2.0 mm in the mesial-distal and 2.5 in the occlusal-cervical and - bucco-lingual directions.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
The restoration survival (changes from baseline up to 36 months) | The treatments will be evaluated after 1 week up to 36 months
  The treatments will be classified "success" when they present clinical satisfactory aspect, and the failures will be scored as "minor failures" and "major failures" (adapted from Innes et al., 2007). The minor failures will be those in which there is a defect in the restoration / crown, but it does not interfere with the tooth health. The major failures will be considered when there signs or symptoms of irreversible pulp damage, such as dental fistula / abscess, tooth fracture or failures that cannot be repaired .The ART-restorations and HT scored as satisfactory will be considered as "successful", while those presented minor and major failures will be considered as "failure".

SECONDARY OUTCOMES:
Child self-reported discomfort | Baseline
  For the assessment of discomfort, the Wong-Baker FACES pain rating scale will be used (Wong; Baker, 1988), which is an ordinal six-point scale ranging from 0 to 5. A score of 0 shows a smiling face, indicating no discomfort, whereas a score of 5 shows a crying and sad face, indicating great discomfort. This method was previously validated for the assessment of pain and discomfort in children (Wong; Baker, 1988; Luffy; Grove, 2003; Novaes et al., 2010)
Perception and concerns related to tooth appearance. | baseline up to 6 months
  The Child's and Parent's Questionnaire about Teeth Appearance will be applied as interview to children in the school as well as being filled out by their parents / caregivers at home (Furtado et al., 2012).
  This instrument has a version for kids and a version for their parents, including questions related to physical, psychological and social order, beyond the perceptions of color change and other aesthetic conditions related to the child´s teeth.
Acceptance of children in relation to treatments performed. | Immediately after treatment (in the same appointment)
  The questionnaire for the evaluation of acceptance in relation to treatment performed will be applied as interview to children in the school. The questionnaire for the children contains 6 items and employs a 5-point pictorial Likert scale. The response possibilities were: strongly agree, agree, indifferent, disagree and strongly disagree. The questionnaires were based on questionnaires used by Bell et al. (2010) They were rewritten in order to be useful for both the ART and the HT. The questionnaires will be translated from English to Portuguese by a Brazilian dentist who is fluent in both languages. The first and last question for the children was identical to control the reliability of answering.
Acceptance of parents in relation to treatments performed. | Immediately after treatment (in the same appointment)
  The questionnaire for the evaluation of acceptance in relation to treatment performed will be filled out by their parents / caregivers at home. The questionnaire for the children contains 6 items and employs a 5-point pictorial Likert scale. The response possibilities were: strongly agree, agree, indifferent, disagree and strongly disagree. The questionnaires were based on questionnaires used by Bell et al. (2010) They were rewritten in order to be useful for both the ART and the HT. The questionnaires will be translated from English to Portuguese by a Brazilian dentist who is fluent in both languages. The first and last question for the children was identical to control the reliability of answering.
Occlusal vertical dimension assessment | The measurements will be done before treatment, immediately after treatment (in the same appointment) and at each check-up appointment (1, 2 and 3 weeks and 1, 6, 12, 18, 24, 30 and 36 months)
  The distance between the most coronal points of the primary canines at the treatment side will be used as determination of the Occlusal vertical dimension assessment (OVD - van der Zee, van Amerongen, 2011).
  The most coronal point of the upper canine will be marked on the lower canine when biting in maximal occlusion using a pencil.
  Subsequently the distance between the marked point and the most coronal point of the lower canine will be measured using a digital calliper (GT-DC-02, Globotronics, Meer, BE). If measuring the OVD score on the treatment side is impossible because of tooth loss, the contralateral side will be used to measure the OVD score.
Cost-effectiveness assessment | Up 36 months
  The cost of treatments will be calculated then taking into account:
  Capital cost: Fixed cost of equipment and instruments such as the cost of autoclave, examination kits; Materials cost or cost of expendable supplies such as gloves, masks, articulating paper, restorative material and PMCs; Labor costs will include salaries of personnel such as a dentist and a dental nurse per day using the maximum levels of the Brazilian Public Health Service salary scales for these professionals in the city treatments will be performed and Time taken to do each procedure of restorative treatments using a stopwatch that will be started when the patient has his/her mouth open and the operator is about to start the restorative intervention and will be stopped when the child stands up from the treatment table.
Oral Health Quality of life (OHRQoL) assessment | Before the treatment and during the 6 months recall
  The perceptions of parents and children regarding the OHRQoL will be evaluated. For that, the Child Perceptions Questionnaire validated for Brazilian children which takes into account the cognitive abilities and lifestyles in an age ranging from 8 to 10 years (CPQ8-10) will be used (Barbosa et al., 2009).
  The instrument consists of 14 questions, distributed into four domains (child symptoms, function, psychological, and self-image/social interaction domains) and in a family impact section (oral symptoms, functional limitations, emotional well-being and social well-being).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Professor, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbosa TS, Tureli MC, Gaviao MB. Validity and reliability of the Child Perceptions Questionnaires applied in Brazilian children. BMC Oral Health. 2009 May 18;9:13. doi: 10.1186/1472-6831-9-13. PMID 19450254
- [Background] Barbosa Tde S, Gaviao MB. Validation of the Parental-Caregiver Perceptions Questionnaire: agreement between parental and child reports. J Public Health Dent. 2015 Fall;75(4):255-64. doi: 10.1111/j.1752-7325.2012.00371.x. Epub 2012 Sep 21. PMID 22994794
- [Background] Bell SJ, Morgan AG, Marshman Z, Rodd HD. Child and parental acceptance of preformed metal crowns. Eur Arch Paediatr Dent. 2010 Oct;11(5):218-24. doi: 10.1007/BF03262750. PMID 20932394
- [Background] Benderli Y, Ulukapi H, Balkanli O, Kulekci G. In vitro plaque formation on some dental filling materials. J Oral Rehabil. 1997 Jan;24(1):80-3. doi: 10.1046/j.1365-2842.1997.00425.x. PMID 9049925
- [Background] Bonifacio CC, Hesse D, Raggio DP, Bonecker M, van Loveren C, van Amerongen WE. The effect of GIC-brand on the survival rate of proximal-ART restorations. Int J Paediatr Dent. 2013 Jul;23(4):251-8. doi: 10.1111/j.1365-263X.2012.01259.x. Epub 2012 Aug 14. PMID 22891625
- [Background] Brito CR, Velasco LG, Bonini GA, Imparato JC, Raggio DP. Glass ionomer cement hardness after different materials for surface protection. J Biomed Mater Res A. 2010 Apr;93(1):243-6. doi: 10.1002/jbm.a.32524. PMID 19557791
- [Background] Carvalho TS, Ribeiro TR, Bonecker M, Pinheiro EC, Colares V. The atraumatic restorative treatment approach: an "atraumatic" alternative. Med Oral Patol Oral Cir Bucal. 2009 Dec 1;14(12):e668-73. PMID 19680186
- [Background] da Mata C, Allen PF, Cronin M, O'Mahony D, McKenna G, Woods N. Cost-effectiveness of ART restorations in elderly adults: a randomized clinical trial. Community Dent Oral Epidemiol. 2014 Feb;42(1):79-87. doi: 10.1111/cdoe.12066. Epub 2013 Aug 19. PMID 23952107
- [Background] de Amorim RG, Leal SC, Frencken JE. Survival of atraumatic restorative treatment (ART) sealants and restorations: a meta-analysis. Clin Oral Investig. 2012 Apr;16(2):429-41. doi: 10.1007/s00784-011-0513-3. Epub 2011 Jan 28. PMID 21274581
- [Background] Fayle SA. UK National Clinical Guidelines in Paediatric Dentistry. Stainless steel preformed crowns for primary molars. Faculty of Dental Surgery, Royal College of Surgeons. Int J Paediatr Dent. 1999 Dec;9(4):311-4. doi: 10.1046/j.1365-263x.1999.00153.x. No abstract available. PMID 10815591
- [Background] Frencken JE, Pilot T, Songpaisan Y, Phantumvanit P. Atraumatic restorative treatment (ART): rationale, technique, and development. J Public Health Dent. 1996;56(3 Spec No):135-40; discussion 161-3. doi: 10.1111/j.1752-7325.1996.tb02423.x. PMID 8915958
- [Background] Frencken JE, Van 't Hof MA, Van Amerongen WE, Holmgren CJ. Effectiveness of single-surface ART restorations in the permanent dentition: a meta-analysis. J Dent Res. 2004 Feb;83(2):120-3. doi: 10.1177/154405910408300207. PMID 14742648
- [Background] Frencken JE, Leal SC, Navarro MF. Twenty-five-year atraumatic restorative treatment (ART) approach: a comprehensive overview. Clin Oral Investig. 2012 Oct;16(5):1337-46. doi: 10.1007/s00784-012-0783-4. Epub 2012 Jul 24. PMID 22824915
- [Background] Gaskin EB, Harless JD, Wefel JS, Guzman-Armstrong S, Armstrong SR, Vargas MA, Hernandez MM, Qian F. Fluorescence changes in remineralized and nonremineralized enamel adjacent to glass ionomer ART restorations: an in vitro study. J Dent Child (Chic). 2007 Sep-Dec;74(3):215-20. PMID 18482517
- [Background] Hesse D, Bonifacio CC, Mendes FM, Braga MM, Imparato JC, Raggio DP. Sealing versus partial caries removal in primary molars: a randomized clinical trial. BMC Oral Health. 2014 May 28;14:58. doi: 10.1186/1472-6831-14-58. PMID 24884684
- [Background] Holmgren CJ, Lo EC, Hu D, Wan H. ART restorations and sealants placed in Chinese school children--results after three years. Community Dent Oral Epidemiol. 2000 Aug;28(4):314-20. doi: 10.1034/j.1600-0528.2000.280410.x. PMID 10901411
- [Background] Holmgren CJ, Roux D, Domejean S. Minimal intervention dentistry: part 5. Atraumatic restorative treatment (ART)--a minimum intervention and minimally invasive approach for the management of dental caries. Br Dent J. 2013 Jan;214(1):11-8. doi: 10.1038/sj.bdj.2012.1175. PMID 23306489
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] Innes NP, Evans DJ, Stirrups DR. Sealing caries in primary molars: randomized control trial, 5-year results. J Dent Res. 2011 Dec;90(12):1405-10. doi: 10.1177/0022034511422064. Epub 2011 Sep 15. PMID 21921249
- [Background] Kandiah T, Johnson J, Fayle SA; British Society of Paediatric Dentistry. British Society of Paediatric Dentistry: a policy document on management of caries in the primary dentition. Int J Paediatr Dent. 2010 Nov;20 Suppl 1:5. doi: 10.1111/j.1365-263X.2010.01087.x. No abstract available. PMID 20718879
- [Background] Kindelan SA, Day P, Nichol R, Willmott N, Fayle SA; British Society of Paediatric Dentistry. UK National Clinical Guidelines in Paediatric Dentistry: stainless steel preformed crowns for primary molars. Int J Paediatr Dent. 2008 Nov;18 Suppl 1:20-8. doi: 10.1111/j.1365-263X.2008.00935.x. PMID 18808544
- [Background] Kornman KS, Loe H. The role of local factors in the etiology of periodontal diseases. Periodontol 2000. 1993 Jun;2:83-97. doi: 10.1111/j.1600-0757.1993.tb00222.x. No abstract available. PMID 9673183
- [Background] Lo EC, Holmgren CJ. Provision of Atraumatic Restorative Treatment (ART) restorations to Chinese pre-school children--a 30-month evaluation. Int J Paediatr Dent. 2001 Jan;11(1):3-10. doi: 10.1046/j.1365-263x.2001.00232.x. PMID 11309870
- [Background] Loe H, Von der Fehr FR, Schiott CR. Inhibition of experimental caries by plaque prevention. The effect of chlorhexidine mouthrinses. Scand J Dent Res. 1972;80(1):1-9. doi: 10.1111/j.1600-0722.1972.tb00257.x. No abstract available. PMID 4502580
- [Background] Luffy R, Grove SK. Examining the validity, reliability, and preference of three pediatric pain measurement tools in African-American children. Pediatr Nurs. 2003 Jan-Feb;29(1):54-9. PMID 12630508
- [Background] Mickenautsch S, Rudolph MJ, Ogunbodede EO, Frencken JE. The impact of the ART approach on the treatment profile in a mobile dental system (MDS) in South Africa. Int Dent J. 1999 Jun;49(3):132-8. doi: 10.1002/j.1875-595x.1999.tb00897.x. PMID 10858745
- [Background] Mickenautsch S, Yengopal V, Banerjee A. Atraumatic restorative treatment versus amalgam restoration longevity: a systematic review. Clin Oral Investig. 2010 Jun;14(3):233-40. doi: 10.1007/s00784-009-0335-8. Epub 2009 Aug 18. PMID 19688227
- [Background] Novaes TF, Matos R, Raggio DP, Imparato JC, Braga MM, Mendes FM. Influence of the discomfort reported by children on the performance of approximal caries detection methods. Caries Res. 2010;44(5):465-71. doi: 10.1159/000320266. Epub 2010 Sep 23. PMID 20861630
- [Background] Paula JS, Torres LH, Ambrosano GM, Mialhe FL. Association between oral health-related quality of life and atraumatic restorative treatment in school children: an exploratory study. Indian J Dent Res. 2012 Nov-Dec;23(6):738-41. doi: 10.4103/0970-9290.111249. PMID 23649055
- [Background] Petersen PE, Bourgeois D, Ogawa H, Estupinan-Day S, Ndiaye C. The global burden of oral diseases and risks to oral health. Bull World Health Organ. 2005 Sep;83(9):661-9. Epub 2005 Sep 30. PMID 16211157
- [Background] Pilot T. Introduction--ART from a global perspective. Community Dent Oral Epidemiol. 1999 Dec;27(6):421-2. doi: 10.1111/j.1600-0528.1999.tb02042.x. No abstract available. PMID 10600075
- [Background] Phantumvanit P, Songpaisan Y, Pilot T, Frencken JE. Atraumatic restorative treatment (ART): a three-year community field trial in Thailand--survival of one-surface restorations in the permanent dentition. J Public Health Dent. 1996;56(3 Spec No):141-5; discussion 161-3. doi: 10.1111/j.1752-7325.1996.tb02424.x. PMID 8915959
- [Background] Raggio DP, Hesse D, Lenzi TL, Guglielmi CA, Braga MM. Is Atraumatic restorative treatment an option for restoring occlusoproximal caries lesions in primary teeth? A systematic review and meta-analysis. Int J Paediatr Dent. 2013 Nov;23(6):435-43. doi: 10.1111/ipd.12013. Epub 2012 Nov 28. PMID 23190278
- [Background] Randall RC, Vrijhoef MM, Wilson NH. Efficacy of preformed metal crowns vs. amalgam restorations in primary molars: a systematic review. J Am Dent Assoc. 2000 Mar;131(3):337-43. doi: 10.14219/jada.archive.2000.0177. PMID 10715925
- [Background] Ricketts D, Lamont T, Innes NP, Kidd E, Clarkson JE. Operative caries management in adults and children. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD003808. doi: 10.1002/14651858.CD003808.pub3. PMID 23543523
- [Background] Roberts JF, Attari N, Sherriff M. The survival of resin modified glass ionomer and stainless steel crown restorations in primary molars, placed in a specialist paediatric dental practice. Br Dent J. 2005 Apr 9;198(7):427-31. doi: 10.1038/sj.bdj.4812197. PMID 15870802
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Splieth CH. Caries management strategies for primary molars: 1-yr randomized control trial results. J Dent Res. 2014 Nov;93(11):1062-9. doi: 10.1177/0022034514550717. Epub 2014 Sep 12. PMID 25216660
- [Background] Santamaria RM, Innes NP, Machiulskiene V, Evans DJ, Alkilzy M, Splieth CH. Acceptability of different caries management methods for primary molars in a RCT. Int J Paediatr Dent. 2015 Jan;25(1):9-17. doi: 10.1111/ipd.12097. Epub 2014 Mar 7. PMID 24602167
- [Background] Schriks MC, van Amerongen WE. Atraumatic perspectives of ART: psychological and physiological aspects of treatment with and without rotary instruments. Community Dent Oral Epidemiol. 2003 Feb;31(1):15-20. doi: 10.1034/j.1600-0528.2003.00021.x. PMID 12542428
- [Background] Schwendicke F, Meyer-Lueckel H, Dorfer C, Paris S. Failure of incompletely excavated teeth--a systematic review. J Dent. 2013 Jul;41(7):569-80. doi: 10.1016/j.jdent.2013.05.004. Epub 2013 May 15. PMID 23685036
- [Background] Svanberg M, Mjor IA, Orstavik D. Mutans streptococci in plaque from margins of amalgam, composite, and glass-ionomer restorations. J Dent Res. 1990 Mar;69(3):861-4. doi: 10.1177/00220345900690030601. PMID 2109000
- [Background] Tay FR, Smales RJ, Ngo H, Wei SH, Pashley DH. Effect of different conditioning protocols on adhesion of a GIC to dentin. J Adhes Dent. 2001 Summer;3(2):153-67. PMID 11570684
- [Background] Tedesco TK, Bonifacio CC, Calvo AF, Gimenez T, Braga MM, Raggio DP. Caries lesion prevention and arrestment in approximal surfaces in contact with glass ionomer cement restorations - A systematic review and meta-analysis. Int J Paediatr Dent. 2016 May;26(3):161-72. doi: 10.1111/ipd.12174. Epub 2015 Jun 12. PMID 26072946
- [Background] van der Zee V, van Amerongen WE. Short communication: Influence of preformed metal crowns (Hall technique) on the occlusal vertical dimension in the primary dentition. Eur Arch Paediatr Dent. 2010 Oct;11(5):225-7. doi: 10.1007/BF03262751. PMID 20932395
- [Background] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Derived] de Araujo MP, Garbim JR, Innes NP, Hesse D, Bonifacio CC, Olegario IC, Braga MM, Mendes FM, Raggio DP. Economic Evaluation of ART and Hall in Primary Molars. BMC Oral Health. 2025 Aug 19;25(1):1336. doi: 10.1186/s12903-025-06528-8. PMID 40830451
- [Derived] Araujo MP, Innes NP, Bonifacio CC, Hesse D, Olegario IC, Mendes FM, Raggio DP. Atraumatic restorative treatment compared to the Hall Technique for occluso-proximal carious lesions in primary molars; 36-month follow-up of a randomised control trial in a school setting. BMC Oral Health. 2020 Nov 11;20(1):318. doi: 10.1186/s12903-020-01298-x. PMID 33176756
- [Derived] Hesse D, de Araujo MP, Olegario IC, Innes N, Raggio DP, Bonifacio CC. Atraumatic Restorative Treatment compared to the Hall Technique for occluso-proximal cavities in primary molars: study protocol for a randomized controlled trial. Trials. 2016 Mar 31;17:169. doi: 10.1186/s13063-016-1270-z. PMID 27029801